CLINICAL TRIAL: NCT02171741
Title: A Phase I Dose Escalation Trial of BIBW 2992 Administration for 20, 13 or 6 Days in Combination With Docetaxel Every 21 Days
Brief Title: Dose Escalation Trial of BIBW 2992 Administration in Combination With Docetaxel in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.6
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib; Docetaxel

ARMS (1):
- Docetaxel + BIBW 2992 (Experimental)
  Interventions: Drug: BIBW 2992; Drug: Docetaxel

INTERVENTIONS:
Drug: BIBW 2992 — continuous daily dosing for 20 or 13 days
Drug: Docetaxel — single infusion on day 1

SUMMARY:
Study to determine the maximum tolerated dose (MTD) for various treatment durations of BIBW 2992 when administered in combination with docetaxel as determined by drug-related adverse events (AEs) as well as Pharmacokinetics, overall safety and antitumor efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with confirmed diagnosis of advanced, non-resectable and / or metastatic solid tumors, of types historically known to express EGFR and/or HER2, who are amenable to docetaxel, preferably patients with breast, prostate, or non-small cell lung cancer. Patients must have failed prior standard therapies associated with clinical benefits, including survival benefits, if such therapies are available. If docetaxel administration is standard therapy associated with clinical benefits, patients are eligible
* Age 18 years or older
* Life expectancy of at least three (3) months
* Written informed consent that is consistent with International Conference on Harmonization - Good Clinical Practice guidelines
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
* Patients must have resolution from prior chemo-, hormone-, immuno-, or radiotherapy related toxicities to CTC Grade <= 1or baseline for individual patient
* Patients must be recovered from previous surgery

Exclusion Criteria:

* Active infectious disease
* Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least eight weeks, no history of cerebral edema or bleeding in the past eight weeks and no requirement for steroids or anti-epileptic therapy
* Cardiac left ventricular function with resting ejection fraction ≥ CTC Grade 1
* Absolute neutrophil count (ANC) less than 1500 / mm3
* Platelet count less than 100 000 / mm3
* Bilirubin > upper limit of normal (ULN)
* Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) > 1.5 x ULN
* Alkaline Phosphatase > 2.5 x ULN
* Serum creatinine > 1.5 mg / dl (> 132 μmol / L, SI (Système Internationale) unit equivalent)
* Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breast-feeding
* Concurrent treatment with other investigational drugs, or chemotherapy, immunotherapy, radiotherapy or hormone therapy (excluding Luteinizing hormone-releasing hormone agonists, or other hormones taken for breast cancer, or bisphosphonates) or participation in another clinical study within the past four weeks before start of therapy or concomitantly with this study
* Treatment with an EGFR- or HER2 inhibiting drug within the past four weeks before start of therapy or concomitantly with this study (8 weeks for trastuzumab)
* Patients unable to comply with the protocol
* Active alcohol or drug abuse
* Hypersensitivity to docetaxel or any component or other drug formulated with polysorbate 80

The patient may be eligible for re-treatment after the previous course is finished. The patient will not be eligible if any of the following conditions are met:

* If patients' latest X-ray, CT or MRI reveals progressive disease, or if clinical assessment reveals signs of disease progression
* Cardiac left ventricular function CTC Grade ≥ 2 at any time during the previous course
* Patients fulfilling any of the Exclusion Criteria listed before as determined before treatment Day 1 of any new course
* Patient not recovered from any dose-limiting toxicity (DLT) 14 days after onset. Recovery is defined as a return to baseline level or CTC Grade 1, whichever is higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence and intensity of AdverseEvents according to Common Terminology Criteria (CTCAE version 3) | up to 32 months
Maximum tolerated dose (MTD) of BIBW 2992 | up to 126 days

SECONDARY OUTCOMES:
Objective tumor response | up to 32 months
Correlation of EGFR (epidermal growth factor receptor), HER2, estrogen receptor (ER) and progesterone receptor (PrR) immunohistochemical status as based on tumor biopsies, or excisions obtained prior to this trial, with objective tumor responses | up to 32 months
Area under the plasma concentration-time curve (AUC) for several time points | up to 48 hours after administration
The percentage of AUC0-∞ that is obtained by extrapolation (%AUCtz-∞) | up to 48 hours after administration
Predose plasma concentration (Cpre) for several time points | predose on day 10 and 21
Plasma concentration at 24 hours (C24) | 24 hours after the first and the last adminstration of study drug
Maximum measured plasma concentration (Cmax) for several time points | up to 48 hours after administration
Time from dosing to the maximum plasma concentration (tmax) for several time points | up to 48 hours after administration
Terminal half-life (t1/2) for several time points | up to 48 hours after administration
Mean residence time (MRT) for several time points | up to 48 hours after administration
Apparent clearance (CL/F) for several timt points | up to 48 hours after administration
Apparent volume of distribution during the terminal phase (Vz/F) for several time points | up to 48 hours after administration
Terminal rate constant in plasma (λz) | up to 48 hours after administration
Accumulation ratio between day 1 and day 21 with respect to Cmax (Ra1) and AUC (RA2) | up to day 21